CLINICAL TRIAL: NCT06401213
Title: MTX-463-I101: A Phase 1 Randomized, Double-Blind, Dose-Escalating Study to Assess the Safety, Tolerability, and Pharmacokinetics of MTX-463 in Healthy Adults
Brief Title: A First-in-Human Safety Trial of MTX-463
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mediar Therapeutics (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MTX-463-I101
Record Dates: First submitted 2024-04-22; First posted 2024-05-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: HEALTHY VOLUNTEER; SAD; MAD; MTX-463-I101; MTX-463; WISP-1; ADULT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTX-463 (Experimental)
  Interventions: Biological: MTX-463
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MTX-463 — MTX-463 is an immunoglobin G1 (IgG1) monoclonal antibody directed against WNT-inducible signaling pathway protein 1 (WISP1). WISP1 (aka CCN-4) is a matricellular protein that appears to be upregulated locally in response to certain chronic diseases and malignancies.
  Arms: MTX-463
Other: Placebo — Matching Placebo-- Normal Saline
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety, tolerability, and PK of single and multiple ascending doses of MTX-463 administered in healthy adults.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety, tolerability, and PK of single and multiple ascending doses of MTX-463 administered in healthy adults.

SAD Portion

The SAD portion of the study will consist of 4 planned dosing cohorts each comprising 8 healthy participants. The starting dose will be 4 mg/kg (Cohort 1) with subsequent planned doses of 8 mg/kg (Cohort 2), 16 mg/kg (Cohort 3), and 30 mg/kg (Cohort 4). Planned doses may be adjusted in response to the data. Additional participants and/or additional dosing cohorts may be added as needed based on the data.

Within each cohort, participants will be randomly assigned to receive MTX-463 or matched placebo. The first 2 participants (sentinel participants) within each cohort will be randomized 1:1 to receive MTX-463 or placebo on Day 1. These participants will be monitored for 24 hours, and after review of the safety data from both participants and approval by the study Investigator and Sponsor's responsible medical officer (SRMO), the additional 6 participants will be randomized to study drug (n=5 MTX-463; n=1 placebo).

Each participant will undergo assessments at specified timepoints on Days 1 through 60. End-of-Study (EOS) procedures will be completed on Day 28 or upon early termination (ET). An End-of-Follow-up (EOF) assessment of PK and ADA will be completed on Day 60.

MAD Portion

The MAD portion of the study will consist of 3 planned dosing cohorts. Each cohort will comprise 8 healthy participants (n=6 MTX-463; n=2 placebo). The starting dose will be a 6.6 mg/kg loading dose and 4 mg/kg maintenance doses (Cohort 1) with subsequent planned doses of a 13 mg/kg loading dose and 8 mg/kg maintenance doses (Cohort 2), and a 27 mg/kg loading dose and 16 mg/kg maintenance doses (Cohort 3). Planned doses may be adjusted in response to the data. Additional participants and/or additional dosing cohorts may be added as needed based on the data.

On Day 1, participants will be randomized to receive either MTX-463 or matched placebo. The randomized participants will receive a single loading dose on Day 1 followed by 2 maintenance doses of study drug on Day 8 and Day 22. Participants will be housed inpatient from Day -1 through post-dose observation on Day 8 and from Day 21 through assessments on Day 29. All other visits will be conducted in the outpatient setting. Each participant will undergo assessments at specified timepoints on Days 1 through 82. End-of-study procedures will be completed on Day 50, or upon ET. An EOF assessment of PK and ADA will be completed on Day 82.

Safety and tolerability of MTX-463 will be reviewed through Day 29 by the study Investigator and SRMO to inform dose escalation decisions for the next dose cohort.

Additional cohorts for the SAD and MAD portions of the study may be added as needed to potentially explore lower doses.

ELIGIBILITY:
Key Inclusion Criteria:

* All genders, ages 18 to 60 years, inclusive
* Willing and able to complete all protocol-required study visits and procedures
* Non-smoker and has not used nicotine- or cotinine-containing products (including tobacco, nicotine gum, patches, and e-cigarettes) for at least 90 days before Screening and until the last study visit
* Willing to refrain from marijuana- or cannabinol-containing products for 90 days before Screening and until the last study visit
* Willing to refrain from ingestion of alcohol from 7 days before Screening until the last study visit
* Agree to a highly effective method of contraception for 28 days prior to the first dose of study drug, and persist through 28 days after the last dose of study drug

Key Exclusion Criteria:

* - Any history of clinically significant lung disease as determined by the Investigator, including but not limited to asthma, chronic obstructive pulmonary disease, pulmonary fibrosis, pulmonary embolus, or pulmonary arterial hypertension
* Any other concurrent active medical condition determined clinically significant by the Investigator
* Body mass index (BMI) >40 kg/m2
* Use of any systemic immunosuppressant medications, medications to treat diabetes, antipsychotics, anticoagulants, or other medications within 90 days of Screening
* Cancer or a history of cancer or lymphoproliferative disorder within 5 years of Screening other than adequately treated non-melanomatous skin cancers or cervical carcinoma in situ
* Current infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) as evidenced by a positive hepatitis B-surface antigen or a positive HIV test at Screening
* Currently pregnant, lactating, or planning to conceive or contribute to pregnancy during the trial and up to 28 days after the participant's last dose of study drug, if applicable
* History of severe depression, psychosis, or suicidal ideation within 5 years of Screening
* History of substance use disorder as specified in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, within 1 year of Screening
* Any clinically significant disease or laboratory abnormality detected at Screening that might interfere with a participant's ability to complete the study, on-study evaluations, or participant safety
* Any surgical procedure, including planned procedures within 12 weeks of Screening
* Participation in another research study of an investigational agent within 30 days of Screening or 5 half-lives of the agent, whichever is longer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events in healthy volunteers | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  Clinical Safety Labs are collected, and Adverse Events are assessed in both inpatient and outpatient clinic visits
MTX-463 PK by dose will be evaluated for Cmax, as feasible | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study
Serum sample results will be summarized for presence of Anti-Drug Antibodies during the SAD and MAD portions of the study. | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study to assess for the presence and titer (if applicable) of Anti-Drug Antibodies.
MTX-463 PK by dose will be evaluated for AUC0-t, as feasible. | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study
MTX-463 PK by dose will be evaluated for AUC0-tau (MAD only), as feasible | Through Day 82 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study
MTX-463 PK by dose will be evaluated for AUC0-∞, as feasible | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  Blood serum samples will be collected at protocol-specified timepoints throughout the study

SECONDARY OUTCOMES:
Blood serum samples will be collected to determine the level of WISP1 engagement of MTX-463 in healthy adult participants | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  These assessments will be summarized as:
  * Change from Baseline in total WISP1 levels
  * Change from Baseline in free WISP1 levels
To assess the effect of baseline body mass index (BMI) on total and free WISP1 levels | Through Day 60 (SAD Cohort) or Day 82 (MAD Cohort)
  Baseline levels and change from Baseline of the total and free WISP1 levels will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.

OTHER OUTCOMES:
To assess the effect of MTX-463 on PD biomarker PRO-C3 for fibrosis in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in fibrosis biomarker PRO-C3 will be evaluated.
To assess the effect of MTX-463 on PD biomarker PRO-C6 for fibrosis in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in fibrosis biomarker PRO-C6 will be evaluated.
To assess the effect of MTX-463 on PD biomarker C7M for fibrosis in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in fibrosis biomarker C7M will be evaluated.
To assess the effect of baseline BMI on PD biomarker IFN-γ for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IFN-γ for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-1β for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-1β for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-2 for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-2 for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-4 for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-4 for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-6 for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-6 for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-10 for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-10 for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-12p70 for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-12p70 for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker IL-17A for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker IL-17A for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker TNF-α for inflammation | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker TNF-α for inflammation will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of MTX-463 on PD biomarker IFN-γ for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IFN-γ will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-1β for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-1β will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-2 for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-2 will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-4 for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-4 will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-6 for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-6 will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-10 for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-10 will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-12p70 for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-12p70 will be evaluated.
To assess the effect of MTX-463 on PD biomarker IL-17A for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker IL-17A will be evaluated.
To assess the effect of MTX-463 on PD biomarker TNF-α for inflammation in healthy adult participants | Through Day 36 (MAD Cohort)
  Change from Baseline in pro-inflammatory biomarker TNF-α will be evaluated.
To assess the effect of baseline BMI on PD biomarker PRO-C3 for fibrosis | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker PRO-C3 for fibrosis will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker PRO-C6 for fibrosis | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker PRO-C6 for fibrosis will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.
To assess the effect of baseline BMI on PD biomarker C7M for fibrosis | Through Day 36 (MAD Cohort)
  Baseline levels and change from Baseline of PD biomarker C7M for fibrosis will be compared in those with BMIs ≥30 kg/m2 to those with BMIs <30 kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Ahad Sabet, MD, Principal Investigator — ICON plc; Jeffrey Bornstein, MD, Study Director — Mediar Therapeutics
Locations (1):
- ICON, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No